CLINICAL TRIAL: NCT06910748
Title: E-training for Medical Professionals On Wellbeing and Effective Resolutions (E.M.P.O.W.E.R.) - A Randomized Controlled Trial
Brief Title: An Internet-based Self-help Intervention to Improve Common Mental Health Problems Among Medical Professionals
Acronym: EMPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Xue YANG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1007627352
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Depression, Anxiety
Keywords: randomized controlled trial; medical professionals; internet-based; self-help; intervention; mental health; depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The EMPOWER program (Experimental): The intervention group will receive 4 weekly sessions (the EMPOWER program) in addition to the information about mental health, depression, anxiety and available treatment and community resources received by the waitlist control group.
  Interventions: Behavioral: E-training for Medical Professionals On Wellbeing and Effective Resolutions (E.M.P.O.W.E.R.)
- Education materials (Active Comparator): The waitlist control group receive education materials about mental health, depression, anxiety and available treatment and community resources but not the EMPOWER prgoram during the intervention period.
  Interventions: Other: Education Materials

INTERVENTIONS:
Behavioral: E-training for Medical Professionals On Wellbeing and Effective Resolutions (E.M.P.O.W.E.R.) — The EMPOWER programme aims to help participants acquire problem-solving skills adapted into the context of MPs' workplace and daily life to address their work-related, personal, and interpersonal problems, including self-neglect, work-life imbalance, patient communication problems, as well as stress during emerging public health crises. The session elements include video introduction, metaphors, daily examples, and narrative stories with prototype MP characters depicting the targeted problems to demonstrate how the taught problem-solving skills could be applied in a variety of situations. Brief exercise and homework will be assigned after each session and personalized written feedback will be provided.
  Arms: The EMPOWER program
Other: Education Materials — The waitlist control receive education materials covering (1) introduction of mental health problems; (2) signs, symptoms, causes, and consequences of anxiety and depression, and (3) treatment approaches and available community resources.
  Arms: Education materials

SUMMARY:
This randomized controlled trial (RCT) aims to evaluate the effectiveness of an internet-based guided self-help intervention developed based on Problem Solving Therapy, a transdiagnostic low-intensity intervention recommended by the World Health Organization, in improving medical professionals' mental health.

DETAILED DESCRIPTION:
Despite the high prevalence of common mental health problems among medical professionals (MPs), their help-seeking for mental health support is low due to barriers such as lack of time, shortage of mental health professionals, and the belief that mental health is not the priority. Existing interventions are empirically effective but practically challenging to be applied in Hong Kong given the long intervention hours and fixed schedule. New interventions are needed to cater for the unique needs of local MPs.

Objectives: An internet-based guided self-help intervention for MPs, E-training for Medical Professionals On Wellbeing and Effective Resolutions (the EMPOWER program), will be developed based on Problem Solving Therapy (PST), a transdiagnostic low-intensity intervention recommended by the World Health Organization. Targeted at local MPs aged 18-60 with depression and/or anxiety symptoms, the intervention aims to reduce their symptoms through strengthening coping skills for work-related problems. A randomized controlled trial (RCT) will be conducted to evaluate (1) the intervention's efficacy in reducing depression/anxiety compared with wait-list control (WLC); (2) its efficacy in improving the levels of PTSD, well-being, burnout, and work performance versus WLC; (3) the potential mediators/mechanisms explaining any between-group differences.

Method: 120 participants will be recruited online. The EMPOWER group will receive four 30-min self-paced weekly intervention sessions. The WLC will receive the intervention after the study period. Data will be collected at baseline, immediately post-intervention and 1-month follow-up. The group effect will be examined by comparing the mean improvement scores and remission rates on the outcome variables among the two groups. The potential mediation effects of adaptive problem solving strategies between the two groups and the outcomes will also be tested.

Expected outcomes: The investigators expect (1) greater reductions in depression and/or anxiety as well as levels of PTSD, well-being, burnout, and work performance for the EMPOWER group at post-treatment and 1-month follow-up than WLC, and that (2) the EMPOWER program will reduce depression and/or anxiety through enhancement in adaptive problem-solving strategies.

Implications: Findings can help to identify a cost-effective, flexible, and readily accessible mental health intervention for local MPs.

ELIGIBILITY:
Inclusion Criteria:

* (1) being a frontline doctor or nurse working in local public settings;
* (2) at least 18 years of age;
* (3) able to read and understand Chinese;
* (4) have access to the Internet; and
* (5) Patient Health Questionnaire (PHQ-9) and/or Generalized Anxiety Disorder (GAD-7) score>=5, indicating at least mild levels of depression and/or anxiety.

Exclusion Criteria:

* (1) currently taking psychotropic medication; and
* (2) actively suicidal.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline depression immediately after the interventions | immediately after the interventions
  The outcome will be measured by the Patient Health Questionnaire (PHQ) consisting of 9 questions designed to correspond to the 9 diagnostic criteria for major depressive disorder listed in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Items are rated from 0 to 3 according to increased frequency of experiencing difficulties in each area covered. Scores are summed and can range from 0 to 27. Score 10 is often recommended as the cut-off score to detect major depressive disorder. Scores of 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe, and severe depression, respectively. The Chinese version has been validated.
Change from baseline depression 1 month after the interventions | 1 month after the interventions
  The outcome will be measured by the Patient Health Questionnaire (PHQ) consisting of 9 questions designed to correspond to the 9 diagnostic criteria for major depressive disorder listed in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Items are rated from 0 to 3 according to increased frequency of experiencing difficulties in each area covered. Scores are summed and can range from 0 to 27. Score 10 is often recommended as the cut-off score to detect major depressive disorder. Scores of 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe, and severe depression, respectively. The Chinese version has been validated.
Change from baseline anxiety immediately after the interventions | Immediately after the interventions
  The outcome will be measured by the Generalized Anxiety Disorder Scale (GAD), which is a 7-item instrument developed to identify likely cases of generalized anxiety disorder in primary care patients. Items are rated for the last two weeks, using a four-point rating scale for duration from 1 ("not at all") to 5 ("nearly every day"). A score of 10 or greater represents a cut point for identifying cases of generalized anxiety disorder, while cut points of 5, 10, 15, and 20 are interpreted as representing mild, moderate, moderately severe, and severe levels of anxiety. The Chinese version has been validated.
Change from baseline anxiety 1 month after the interventions | 1 month after the interventions
  The outcome will be measured by the Generalized Anxiety Disorder Scale (GAD), which is a 7-item instrument developed to identify likely cases of generalized anxiety disorder in primary care patients. Items are rated for the last two weeks, using a four-point rating scale for duration from 1 ("not at all") to 5 ("nearly every day"). A score of 10 or greater represents a cut point for identifying cases of generalized anxiety disorder, while cut points of 5, 10, 15, and 20 are interpreted as representing mild, moderate, moderately severe, and severe levels of anxiety. The Chinese version has been validated.

CONTACTS AND LOCATIONS:
Locations (1):
- JC School of Public Health and Primary Care, Faculty of Medicine, CUHK, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No